CLINICAL TRIAL: NCT01686152
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Multicenter Study Comparing Imiquimod Cream, 3.75% to Zyclara® (Imiquimod) Cream, 3.75% in the Treatment of Actinic Keratosis of the Face or Balding Scalp
Brief Title: Study Comparing Imiquimod Cream, 3.75% to Zyclara® (Imiquimod) Cream, 3.75% in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SYM 2012-01
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational Test Product (Experimental): Imiquimod Cream, 3.75% (Teva)
  Interventions: Drug: Imiquimod Cream, 3.75%
- Reference Listed Drug (Active Comparator): Zyclara® (imiquimod Cream), 3.75% (Medicis)
  Interventions: Drug: Zyclara®
- Vehicle (Placebo Comparator): Vehicle of Test Product (Teva)
  Interventions: Other: Vehicle of Test Product

INTERVENTIONS:
Drug: Imiquimod Cream, 3.75%
  Arms: Investigational Test Product
Drug: Zyclara®
  Other Names: Imiquimod Cream (generic name)
  Arms: Reference Listed Drug
Other: Vehicle of Test Product
  Arms: Vehicle

SUMMARY:
To determine the comparability of the safety and efficacy of Imiquimod Cream, 3.75% and Zyclara (imiquimod) Cream, 3.75% (the reference listed drug) in subjects with actinic keratosis (AK) of the face or balding scalp. It will also be determined whether the efficacy of each of the two active treatments is superior to that of the Vehicle cream.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the study
* At least 18 years of age.
* Immunocompetent male or non-pregnant and non-lactating female. Each female subject of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years), in addition to having a negative urine pregnancy test at Visit 1/Day 1, must be willing to use an acceptable form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double-barrier methods (for example, condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active. Subjects entering the study who are on hormonal contraceptives (oral contraceptives, patches and injection) must have been on this method for at least 3 months (90 days) prior to the study and continue the method for the duration of the study. Subjects who had used hormonal contraception (oral contraceptives, patches and injection) and stopped must have stopped no less than 3 months (90 days) prior to baseline. Subjects entering the study using contraceptive implants and intrauterine contraceptives must have been on this method for at least 6 months (180 days) and continue for the duration of the study and if they stopped must have stopped no less than 6 months (180 days) prior to baseline.
* Clinical diagnosis of AK, defined as ≥ 5 and ≤ 20 clinically typical, visible or palpable AK lesions, each at least 4 mm in diameter, in an area that exceeds 25 cm2 on either the face (excluding ears) or balding scalp, but not both face and scalp.
* In general good health and free from any clinically significant disease, other than AK, that might interfere with the study evaluations.
* Willing and able to understand and comply with the requirements of the study, apply the IP as instructed, attend the required visits, comply with therapy prohibitions, and be able to complete the study.

Exclusion Criteria:

* Presence of atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, or other possible confounding skin conditions on the treatment area of either the face or balding scalp.
* Clinically significant systemic disease (immunological deficiencies), unstable medical disorder, life-threatening disease, or current malignancies.
* Use on the face or balding scalp of chemical peel, dermabrasion, laser abrasion, psoralen plus ultraviolet A (PUVA) therapy, and/or ultraviolet B (UVB) therapy in the last 6 months (180 days)
* Use of any systemic cancer chemotherapy medications in the last 6 months (180 days)
* Use on the face or balding scalp of cryodestruction or chemodestruction, curettage, photodynamic therapy, surgical excision, topical 5-fluorouracil, topical corticosteroids, topical diclofenac, topical imiquimod, topical retinoids, masoprocol, or other treatments for AK in the last 1 month (30 days)
* Immunomodulators or immunosuppressive therapies, interferon, oral/systemic corticosteroids, or cytotoxic drugs in the last 1 month (30 days). Intranasal or inhaled corticosteroids are acceptable if kept constant throughout the study.
* Need or intent to continue to use any treatment listed in the four points above during the current study
* Known hypersensitivity or allergies to imiquimod or any component of the IP (in any dosage form).
* Females who are pregnant, breastfeeding, intending to become pregnant during the study, or who do not agree to use an acceptable form of birth control during the study.
* Any clinically significant condition or situation other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
* Use of any investigational drug or investigational device within 1 month (30 days) prior to randomization.
* Previous participation in this study.
* Sunburn in the designated treatment area to be treated at study entry.
* Current involvement in activities that require excessive or prolonged sun exposure.
* Consumption of excessive amounts of alcohol, abuse drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Radiant Research, Inc., Tucson, Arizona
  - Encino Research Center, Encino, California
  - Dermatology Research Associates, Los Angeles, California
  - Northern California Research, Sacramento, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Longmont Clinic, PC, Longmont, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Tory Sullivan, M.D., P.A., North Miami Beach, Florida
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Leavitt Medical Associates of Florida dba Ameriderm Research, Ormond Beach, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Dermatology Specialists Research LLC, Louisville, Kentucky
  - Radiant Research, Inc., Cincinnati, Ohio
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Research Across America, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Test Product | Reference Listed Drug | Vehicle
Started | 252 | 253 | 84
Completed | 211 | 218 | 75
Not Completed | 41 | 35 | 9
Not completed — Withdrawal by Subject | 11 | 11 | 3
Not completed — Drug Code Unblinded | 0 | 1 | 0
Not completed — Protocol Violation | 6 | 1 | 0
Not completed — Adverse Event | 12 | 11 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — IP Non-compliance | 5 | 5 | 0
Not completed — Lost to Follow-up | 7 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Safety Population Data Included
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Test Product | Reference Listed Drug | Vehicle | Total
Number analyzed (Participants) | 247 | 249 | 80 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (9.12) | 68.6 (9.79) | 68.7 (10.23) | 68.3 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 27 | 13 | 84
  Male | 203 | 222 | 67 | 492
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 2 | 24
  Not Hispanic or Latino | 237 | 237 | 78 | 552
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 246 | 249 | 80 | 575
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Location of Lesion [Count of Participants; unit: Participants]
  Scalp | 115 | 135 | 35 | 285
  Face | 132 | 114 | 45 | 291
Size (cm^2) of Lesion [Mean (Standard Deviation); unit: cm2] | 317.5 (178.53) | 305.8 (180.78) | 335.7 (183.78) | 315 (180.20)
Number of Visible or Palpable Lesions [Mean (Standard Deviation); unit: lesions] | 10.6 (3.98) | 10.7 (4.16) | 11.0 (4.35) | 10.7 (4.11)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success/Failure at Visit 5/Week 14
Description: The primary efficacy endpoint is the proportion of subjects with treatment success at Visit 5/Week 14 (8 weeks post-treatment). Treatment success is defined as 100% clearance of all AK lesions (baseline AK lesions and any new AK lesions) within the treatment area.
Time Frame: 14 Weeks
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Test Product | Reference Listed Drug | Vehicle
Number analyzed (Participants) | 178 | 179 | 64
Participants
  Success (100% clearance of AK lesions) | 42 | 40 | 6
  Failure <100% clearance of AK lesions | 136 | 139 | 58
Statistical Analysis 1: Comparison: Investigational Test Product vs Reference Listed Drug; Test type: Equivalence — The test product was determined to be bioequivalent to the reference product if the 90% confidence interval was within -0.20 to 0.20; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.0663 to 0.0913]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Investigational Test Product | Reference Listed Drug | Vehicle
All-Cause Mortality (participants affected / at risk) | 1/247 | 0/249 | 0/80
Serious Adverse Events (participants affected / at risk) | 6/247 | 8/249 | 1/80
Other Adverse Events (participants affected / at risk) | 81/247 | 77/249 | 16/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Test Product (N=247) | Reference Listed Drug (N=249) | Vehicle (N=80)
Cerebrovascular accident (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Umbilical Hernia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Laceration (scalp) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis Ischemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic Gastroparesis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Ligament Rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Test Product (N=247) | Reference Listed Drug (N=249) | Vehicle (N=80)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0
Eyelid Oedema (Eye disorders) | 1 | 1 | 0
Lacrimation Increased (Eye disorders) | 1 | 0 | 1
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0
Retinal Tear (Eye disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Colonic Polyp (Gastrointestinal disorders) | 1 | 1 | 0
Diabetic Gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival Inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Lip Erosion (Gastrointestinal disorders) | 1 | 1 | 0
Lip Pain (Gastrointestinal disorders) | 2 | 0 | 0
Lip Swelling (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Application Site Dermatitis (General disorders) | 2 | 0 | 0
Application Site Erythema (General disorders) | 1 | 0 | 0
Application Site Haemorrhage (General disorders) | 1 | 0 | 0
Application Site Pain (General disorders) | 2 | 4 | 0
Application Site Pruritus (General disorders) | 0 | 2 | 0
Application Site Reaction (General disorders) | 0 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 0
Chills (General disorders) | 3 | 2 | 0
Discomfort (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 4 | 0
Influenza Like Illness (General disorders) | 5 | 10 | 0
Local Swelling (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 3 | 1 | 0
Oedema Mucosal (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 0
Tenderness (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Allergy to Arthropod Sting (Immune system disorders) | 0 | 0 | 1
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0
Adenoviral Upper Respiratory Infection (Infections and infestations) | 1 | 0 | 0
Application Site Cellulitis (Infections and infestations) | 1 | 0 | 0
Application Site Infection (Infections and infestations) | 1 | 0 | 0
Bacterial Infections (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Dental Fistula (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 3 | 0
Herpes Zoster (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1
Oral Herpes (Infections and infestations) | 3 | 3 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1
Rash Pustular (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 2 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 5 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skin Injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Superficial Injury of Eye (Injury, poisoning and procedural complications) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 5 | 0
Headache (Nervous system disorders) | 8 | 8 | 1
Lethargy (Nervous system disorders) | 2 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Nightmare (Psychiatric disorders) | 2 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin Erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may not publish results from this generic (ANDA) study unless reviewed and approved by sponsor.